CLINICAL TRIAL: NCT02314169
Title: A Multi-Institutional Phase 2 Study of Nivolumab or Nivolumab in Combination With Ipilimumab in Refractory Metastatic Squamous Cell Carcinoma of the Anal Canal
Brief Title: Nivolumab With or Without Ipilimumab in Treating Patients With Refractory Metastatic Anal Canal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-02420; NCI-2014-02420 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI9673; P9673_R03PAPPHOLD01; 9673 (Other: Yale University Cancer Center LAO); 9673 (Other: CTEP); N01CM00032 (NIH); N01CM00038 (NIH); N01CM00039 (NIH); N01CM00071 (NIH); N01CM00099 (NIH); N01CM00100 (NIH); P30CA016359 (NIH); U10CA180821 (NIH); UM1CA186704 (NIH); UM1CA186712 (NIH); UM1CA186716 (NIH)
Record Dates: First submitted 2014-12-10; First posted 2014-12-11 (Estimated); Last update posted 2025-04-29 (Actual); Status verified 2025-03

CONDITIONS: Anal Canal Squamous Cell Carcinoma; Metastatic Anal Canal Carcinoma; Stage IV Anal Cancer AJCC v8
MeSH Terms: conditions — Anal Canal Carcinoma; Anus Neoplasms | interventions — Specimen Handling; Ipilimumab; CTLA-4 Antigen; Magnetic Resonance Spectroscopy; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A (nivolumab) (Experimental): Patients receive nivolumab IV over 60 minutes once every two weeks. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, MRI and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab
- Part B Arm I (nivolumab) (Experimental): Patients receive nivolumab IV over 30 minutes once every 4 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, MRI and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab
- Part B Arm II (nivolumab, ipilimumab) (Experimental): Patients receive nivolumab as in Arm I. Patients also receive ipilimumab IV over 30 minutes once every 8 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, MRI and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
  Arms: Part B Arm II (nivolumab, ipilimumab)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo

SUMMARY:
This phase II trial studies how well nivolumab with or without ipilimumab works in treating patients with anal canal cancer that has not responded to previous treatment (refractory) and that has spread from where it first started (primary site) to other places in the body (metastatic). Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate overall response rate (ORR) with nivolumab in patients with previously treated metastatic squamous cell carcinoma (SCCA) of the anal canal. (Part A) II. To determine an improvement in progression-free survival (PFS) when nivolumab is combined with ipilimumab versus (vs.) nivolumab alone in patients with previously treated metastatic SCCA (Part B).

SECONDARY OBJECTIVES:

I. To evaluate progression-free survival (PFS) of nivolumab in patients with previously treated metastatic SCCA of the anal canal. (Part A) II. To evaluate overall survival (OS) in patients with previously treated metastatic SCCA of the anal canal treated with nivolumab. (Part A) III. To evaluate the grade 3 and 4 toxicity rate in patients with previously treated metastatic SCCA of the anal canal when treated with nivolumab. (Part A) IV. To evaluate the overall response rate (ORR) of nivolumab plus or minus ipilimumab in patients with previously treated metastatic SCCA of the anal canal. (Part B) V. To evaluate overall survival (OS) in patients with previously treated metastatic SCCA of the anal canal treated with nivolumab plus or minus ipilimumab. (Part B) VI. To evaluate the grade 3 and 4 toxicity rate in patients with previously treated metastatic SCCA of the anal canal when treated with nivolumab plus or minus ipilimumab. (Part B)

EXPLORATORY OBJECTIVES:

I. To evaluate ORR, PFS, and OS based on expression of programmed cell death 1 ligand 1 (PD-L1), programmed cell death 1 (PD-1), peritumoral cluster of differentiation (CD)8+ tumor infiltrating lymphocytes (TILs), peritumoral CD4+ TILs, and regulatory T cells as analyzed from tumor biopsies in previously treated patients with metastatic SCCA of the anal canal when treated with nivolumab. (Part A) II. To evaluate radiographic responses according to relative changes in proportions of anti-human papillomavirus (HPV) specific CD8+ and CD4+ TILs and regulatory T cells in patients with previously treated metastatic SCCA of the anal canal following treatment with nivolumab, analyzed from serial peripheral blood samples. (Part A) III. To evaluate ORR, PFS, and OS based on expression of PD-L1, PD-1, peritumoral CD8+ tumor infiltrating lymphocytes (TILs), peritumoral CD4+ TILs, and regulatory T cells as analyzed from tumor biopsies in previously treated patients with metastatic SCCA of the anal canal when treated with nivolumab plus or minus ipilimumab. (Part B) IV. To evaluate radiographic responses according to relative changes in proportions of anti-HPV specific CD8+ and CD4+ TILs and regulatory T cells in patients with previously treated metastatic SCCA of the anal canal following treatment with nivolumab plus or minus ipilimumab. (Part B)

OUTLINE:

PART A: Patients receive nivolumab intravenously (IV) over 60 minutes once every two weeks. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) scan, magnetic resonance imaging (MRI) and blood sample collection throughout the study.

PART B: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive nivolumab IV over 30 minutes once every 4 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, MRI and blood sample collection throughout the study.

ARM II: Patients receive nivolumab as in Arm I. Patients also receive ipilimumab IV over 30 minutes once every 8 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, MRI and blood sample collection throughout the study.

After completion of study treatment, patients are followed up for 100 days and then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed previously treated metastatic squamous cell carcinoma of the anal canal
* Patients must have measurable disease according to the standard Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. CT scans or MRIs used to assess the measurable disease must have been completed within 28 days prior to study drug initiation
* Patients must have been treated with at least one prior systemic treatment for incurable advanced or metastatic SCCA of the anal canal; prior treatment for metastatic disease is not required for patients who develop new metastatic lesions during or within 6 months of completion of chemoradiation for limited-stage disease; patients who receive chemotherapy for incurable advanced or metastatic SCCA of the anal canal must wait a minimum >= 28 days (6 weeks for nitrosoureas or mitomycin C) after the date of completion of chemotherapy prior to initiating treatment with nivolumab on this study; patients who undergo palliative radiotherapy to a site of tumor must wait a minimum >= 28 days from the date of completion of radiotherapy prior to initiating treatment with nivolumab (Part A and B) or nivolumab +/- Ipilimumab (Part B) on this study
* Patients must be of age >= 18 years at the time of study registration; because no dosing or adverse event data are currently available on the use of nivolumab in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 (Karnofsky >= 80%)
* Leukocytes >= 2,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Hemoglobin >= 9.0 gm/dL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (except patients with Gilbert syndrome, who can have total bilirubin < 3.0 mg/dL)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN
* Serum creatinine =< 1.5 x ULN OR creatinine clearance (CrCl) >= 50 mL/min (if using the Cockcroft-Gault formula)
* Before study enrollment, women of child bearing potential must be advised of the importance of avoiding pregnancy during study participation and the potential risk factors for an unintentional pregnancy; the subject must sign an informed consent form documenting this discussion; the effects of nivolumab and ipilimumab on the developing human fetus are unknown; for this reason women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; women of childbearing potential MUST have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to the start of nivolumab with or without ipilimumab; the minimum sensitivity of the pregnancy test must be 25 IU/L or equivalent units of HCG; if the pregnancy test is positive, the subject must not receive nivolumab with or without ipilimumab and must not be enrolled in the study
* Women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal; menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes
* WOCBP receiving nivolumab (Parts A+B) or nivolumab and ipilimumab (Part B) will be instructed to adhere to contraception for a period of 5 months after the last dose of investigational product; men receiving nivolumab (Parts A+B) or nivolumab and ipilimumab (Part B only) and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of investigational product; these durations have been calculated using the upper limit of the half-life for nivolumab (25 days) and are based on the protocol requirement that WOCBP use contraception for 5 half-lives plus 30 days and men who are sexually active with WOCBP use contraception for 5 half-lives plus 90 days
* Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she (or the participating partner) should inform the treating physician immediately; if, following initiation of the investigational product, it is subsequently discovered that a study subject is pregnant or may have been pregnant at the time of investigational product exposure, including during at least 6 half-lives after product administration, the investigational product will be permanently discontinued in an appropriate manner (e.g., dose tapering if necessary for subject safety); the investigator must immediately notify BMS of this event and record the pregnancy on the Pregnancy Surveillance Form (not an severe adverse event [SAE] form); initial information on a pregnancy must be reported immediately to BMS, and the outcome information provided once the outcome is known; completed Pregnancy Surveillance Forms must be forwarded to BMS according to SAE reporting procedures; any pregnancy that occurs in a female partner of a male study participant should be reported to the sponsor. Information on this pregnancy will be collected on the Pregnancy Surveillance Form; protocol-required procedures for study discontinuation and follow-up must be performed on the subject unless contraindicated by pregnancy (e.g., X-ray studies); other appropriate pregnancy follow-up procedures should be considered if indicated; in addition, the investigator must report and follow-up on information regarding the course of the pregnancy, including perinatal and neonatal outcome; infants should be followed for a minimum of 8 weeks
* Ability to understand and the willingness to sign a written informed consent document
* Brain metastases are allowed if they have been adequately treated with radiotherapy or surgery and have been stable for at least three months prior to registration; eligible subjects should be neurologically asymptomatic; there is no magnetic resonance imaging (MRI) evidence of progression for a minimum of 4 weeks after treatment is complete and within 28 days prior to the first dose of nivolumab administration; there must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration
* Willingness for evaluation of cardiac function including electrocardiography (EKG) and echocardiogram (ECHO) cardiogram for any patients with a history of congestive heart failure (CHF) or at risk because of underlying cardiovascular disease or exposure to cardiotoxic drugs as clinically indicated
* All patients must be willing to undergo testing for human immunodeficiency virus (HIV) testing if not tested within the past 6 months
* If HIV+ positive, all patients infected with human immunodeficiency virus (HIV) may be eligible for study provided that their CD4+ count >= 300/uL; their viral load is undetectable; they are currently receiving highly active antiretroviral therapy (HAART)
* All HIV+ patients will be under the care of an infectious diseases specialist; if a relationship with an infectious diseases specialist is not established, infectious disease specialist will be consulted; records of all viral counts and peripheral T-cell counts must be sent to the study coordinator in order to follow these values over the course of treatment
* All patients must be willing to be tested for hepatitis screening; patients co-infected with hepatitis B virus and/or hepatitis C virus may be included in this study provided that their liver function tests remain within the limits listed above; patients must be followed by a hepatologist during the course of this study

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events (AEs) due to agents administered more than 4 weeks earlier (i.e., grade >= 2 AE present); palliative (limited-field) radiation therapy is permitted, as long as the lesion being considered for palliative radiation is not a target lesion
* Patients who are receiving any other investigational agents
* Patients should be excluded if they have had prior treatment with an anti-PD-1, anti-PD-L1, anti-programmed cell death ligand 2 (PD-L2), anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab (Parts A+ B) and/or ipilimumab (Part B)
* History of severe hypersensitivity reaction to any monoclonal antibody
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including chronic prolonged systemic corticosteroids (defined as corticosteroid use of duration one month or greater), should be excluded; these include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or anti-phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration; inhaled or topical steroids and adrenal replacement doses =< 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease; patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption); physiologic replacement doses of systemic corticosteroids are permitted, even if =< 10 mg/day prednisone equivalents; a brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for at least three years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-05-13 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2026-03-21 (Estimated)

PRIMARY OUTCOMES:
Overall response rate: number of participants with response (Part A) | Up to 2 years
  Responses assessed using computed tomography (CT) scans or magnetic resonance imaging according to standard Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria in order to assess disease progression. Complete Response (CR): Disappearance all target lesions; any pathological lymph nodes reduction in short axis to < 10 mm (< 1 cm). Partial Response (PR): > 30% decrease in sum diameters of target lesions. Progressive Disease (PD): > 20% increase in sum diameters lesions. (Note: appearance of one or > new lesions considered progressions). Stable Disease (SD): Neither shrinkage qualify for PR nor increase for PD.
Progression-free survival (PFS) (Part B) | Time period from the date of randomization to the date of PD or death whichever occurred first, assessed up to 2 years

SECONDARY OUTCOMES:
Number of participants with toxicities (Part A) | Up to 100 days post-treatment
  Will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The most frequent of adverse events measured relative to the total number of patients treated, and the toxicities tabulated by grade according to CTCAE.
Overall survival (Part A and B) | From initiation of treatment with nivolumab until death, assessed up to 2 years
  Time measured from initiation of treatment with nivolumab till death. Kaplan-Meier analysis will be performed to estimate the median overall survival with a 95% confidence interval.
Progression-free Survival (Part A) | From initiation of treatment with nivolumab until the time of disease progression, assessed up to 2 years
  From initiation of treatment with nivolumab until the time of disease progression, time measured in months. Kaplan-Meier analysis performed to estimate the median progression-free survival with a 90% confidence interval.
Overall response rates (Part B) | Up to 2 years
  Responses assessed using CT scans or magnetic resonance imaging according to standard RECIST 1.1 criteria in order to assess disease progression. CR: Disappearance all target lesions; any pathological lymph nodes reduction in short axis to < 10 mm (< 1 cm). PR: > 30% decrease in sum diameters of target lesions. PD: > 20% increase in sum diameters lesions. (Note: appearance of one or > new lesions considered progressions). SD: Neither shrinkage qualify for PR nor increase for PD.
Incidence of grade 3/4/5 adverse events (Part B) | Up to 2 years
  Will be assessed by CTCAE version 5.0.

OTHER OUTCOMES:
Expression of biomarkers using immunohistochemistry and blood samples (Part A) | Up to time of treatment discontinuation
  Descriptive statistics including plots, mean, median and standard deviations will be used to summarize data. For continuous outcomes, t-test and analysis of variance will be used to compare outcome measures across patient characteristics. Pair-wise comparisons will be performed using pre- and post-therapy samples from each patient. The chi-square test or Fisher's exact test will be used to test the association between two categorical variables. Both univariate and multivariate logistic regressions will be performed to model prognostic factors.

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Eng, Principal Investigator — Yale University Cancer Center LAO
Locations (56):
- United States (55):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Morris VK, Salem ME, Nimeiri H, Iqbal S, Singh P, Ciombor K, Polite B, Deming D, Chan E, Wade JL, Xiao L, Bekaii-Saab T, Vence L, Blando J, Mahvash A, Foo WC, Ohaji C, Pasia M, Bland G, Ohinata A, Rogers J, Mehdizadeh A, Banks K, Lanman R, Wolff RA, Streicher H, Allison J, Sharma P, Eng C. Nivolumab for previously treated unresectable metastatic anal cancer (NCI9673): a multicentre, single-arm, phase 2 study. Lancet Oncol. 2017 Apr;18(4):446-453. doi: 10.1016/S1470-2045(17)30104-3. Epub 2017 Feb 18. PMID 28223062